CLINICAL TRIAL: NCT07406737
Title: Feasibility and Outcomes Registry of Lumenless dEfibrillation Leads for Conduction System Pacing
Acronym: FORGE CSP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Pierre OLLITRAULT, MD, University Hospital, Caen
Other Study IDs: 2026-RYTHMO-01
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Resynchronization Therapy; Left Bundle Branch Area Pacing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recent development and market introduction of small diameter implantable defibrillation leads able to deliver left bundle branch area pacing (LBBAP) has opened the possibility of achieving cardiac resynchronization therapy (CRT) using a single- or dual-chamber implantable-cardioverter defibrillator (ICD). This approach may reduce the number of intracardiac leads required and, consequently, has the potential to lower both procedural and long-term complication rates. However, the integration of these leads into currently recommended CRT strategies remains hypothetical. The FORGE CSP registry will prospectively enroll patients with an indication for CRT in whom implantation of a LBBAP ICD lead is attempted.

DETAILED DESCRIPTION:
The FORGE CSP Registry is a prospective, multicentre and nationwide, post-approval registry, including consecutive patients with an indication for CRT and in whom implantation of a LBBAP ICD lead is attempted as a first line strategy.

The primary objective of this registry is to measure the proportion of patients who achieve effective CRT solely through the use of a LBBAP ICD lead (plus right atrial lead if appropriate).

The secondary objectives of this registry are: (1) to assess the feasibility of the LBBAP ICD lead implantation (regarding LBBAP validated electrophysiologic criteria) and the associated learning curve; (2) to evaluate the incidence of implantation of a third lead, namely a left ventricular lead positioned in the coronary sinus, in combination with the LBBAP ICD lead (LOT-CRT); (3) to assess the risk of complications related to the use of the LBBAP ICD lead, including its impact on tricuspid valve function, the risk of lead dislodgement, and other procedure- or device-related complications; (4) to evaluate de cost-effectiveness of CRT using LBBAP ICD lead, compared with conventional CRT; (5) and to compare CRT response in LBBAP ICD lead recipients, versus historical cohort of conventional CRT.

ELIGIBILITY:
Inclusion Criteria:

* age > 18-year-old
* indication for CRT according to current ESC/EHRA guidelines
* first-line LBBAP ICD lead implantation attempted
* national insurance coverage

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a validated CRT indication for whom the implantation of a LBBAP ICD lead in attempted as a first-line strategy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
LBBAP ICD lead CRT efficacy | 0 - 3 Months
  Proportion of patients with an effective CRT (defined by LBBAP validated ECG criteria) using solely the LBBAP ICD lead (plus right atrial lead if appropriate).

SECONDARY OUTCOMES:
LBBAP ICD lead implantation feasibility | Procedural
  Incidence of successful LBBAP ICD lead implantation (defined by LBBAP ECG validated criteria)
LOT-CRT utilization | Procedural
  Incidence of coronary sinus left ventricular lead implantation (in addition to LBBAP ICD lead)
Safety of LBBAP ICD lead | 0 - 3 Months
  Incidence of ICD lead micro or macro-dislodgment Incidence of de novo tricuspid regurgitation (grade > or = 3) Incidence of loss of CRT (based on LBBAP validated ECG criteria)
Cost-effectiveness | Procedural
  Comparaison of device-associated costs in LBBAP ICD lead recipients and conventional CRT recipients.

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vijayaraman P, Liu X, Denman R, Schloss EJ, Whinnett ZI, Kron J, Jastrzebski M, Zakaib JS, Abhayaratna WP, Philippon F, Afzal MR, Pokharel P, Burrell J, Tanner J, Geelen T, Platner ML, Butler K, Mason PK, Crossley GH; LEADR LBBAP Trial Investigators. Safety and performance of a novel defibrillation lead for left bundle branch area placement: Primary results of the LEADR LBBAP clinical trial. Heart Rhythm. 2025 Oct 17:S1547-5271(25)02981-9. doi: 10.1016/j.hrthm.2025.10.028. Online ahead of print. PMID 41110529
- [Background] Crossley GH 3rd, Sanders P, Hansky B, De Filippo P, Shah MJ, Shoda M, Khelae SK, Richardson TD, Philippon F, Zakaib JS, Tse HF, Sholevar DP, Stellbrink C, Pathak RK, Milasinovic G, Chinitz JS, Tsang B, West MB, Ramza BM, Han X, Bozorgnia B, Carta R, Geelen T, Himes AK, Platner ML, Thompson AE, Mason PK; Lead EvaluAtion for Defibrillation and Reliability Trial Investigators. Safety, efficacy, and reliability evaluation ofa novel small-diameter defibrillation lead: Global LEADR pivotal trial results. Heart Rhythm. 2024 Oct;21(10):1914-1922. doi: 10.1016/j.hrthm.2024.04.067. Epub 2024 May 17. PMID 38762820
- [Background] Sanders P, Mason PK, Hansky B, De Filippo P, Shah MJ, Sholevar DP, Zakaib JS, Philippon F, Tsang B, Pathak RK, Richardson TD, Friedman M, Schaller RD, Anguera I, Mihalcz A, Bozorgnia B, Thompson AE, Arias K, Maus B, Bounds C, Crossley GH. Sensing and detection performance of the novel, small-diameter OmniaSecure defibrillation lead: in-depth analysis from the LEADR trial. Europace. 2025 Mar 28;27(4):euaf062. doi: 10.1093/europace/euaf062. PMID 40127675
- [Background] Crossley GH 3rd, Mason PK, Hansky B, De Filippo P, Shah MJ, Philippon F, Sholevar D, Richardson TD, West MB, Dinerman J, Dawson J, Himes A, Severseike L, Thompson AE, Sanders P. High predicted durability for the novel small-diameter OmniaSecure defibrillation lead. Heart Rhythm. 2025 Feb;22(2):302-310. doi: 10.1016/j.hrthm.2024.09.005. Epub 2024 Sep 26. PMID 39341436
- [Background] Crossley GH, Sanders P, Hansky B, De Filippo P, Shah MJ, Khelae SK, Richardson TD, Philippon F, Zakaib JS, Geelen T, Arias K, Maus B, Mason PK; Lead EvaluAtion for Defibrillation and Reliability Trial Investigators. Safety and Efficacy of the Novel OmniaSecure Defibrillation Lead Through Long-Term Follow-Up: Final Results From the LEADR Trial. Circ Arrhythm Electrophysiol. 2026 Jan;19(1):e014424. doi: 10.1161/CIRCEP.125.014424. Epub 2025 Nov 12. PMID 41222500